CLINICAL TRIAL: NCT04880330
Title: Interest of an Auriculotherapy Session in Smoking Cessation Controlled, Randomized, Single-blind Study: Proof of Concept Study
Brief Title: Interest of an Auriculotherapy Session in Smoking Cessation
Acronym: StopAuric
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hopital Foch (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2019_0139
Record Dates: First submitted 2021-05-05; First posted 2021-05-10 (Actual); Last update posted 2024-06-14 (Actual); Status verified 2024-06

CONDITIONS: Tobacco Use Cessation
MeSH Terms: conditions — Tobacco Use Cessation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Cryo-Auriculotherapy (Experimental): Patients benefit from 1 session of cryo-auriculotherapy with device with nitrous oxyde on 15 auricular points.
  Interventions: Device: Cryo-Auriculotherapy
- Sham Comparator: Control group (Sham Comparator): Patients benefit from 1 session of cryo-auriculotherapy with device without nitrous oxyde on 15 auricular points..
  Interventions: Device: Sham comparator

INTERVENTIONS:
Device: Cryo-Auriculotherapy — 1 session of cryo-auriculotherapy with device with nitrous oxyde on 15 auricular points.
  Arms: Experimental: Cryo-Auriculotherapy
Device: Sham comparator — 1 session of cryo-auriculotherapy with device without nitrous oxyde on 15 auricular points.
  Arms: Sham Comparator: Control group

SUMMARY:
The aim of the study is to show that auriculotherapy is effective in smoking cessation.

DETAILED DESCRIPTION:
Smoking is a major risk factor for morbidity and mortality. The French High Authority for Health recommends that "All health professionals must advise every smoker to stop smoking, regardless of the form of tobacco used, and offer advice and assistance to quit". The modalities of accompaniment towards quitting and support during the withdrawal period vary according to each smoker, his or her degree of motivation, the intensity of his or her dependence, and any previous attempts.

Nicotine substitutes are the first-line drug treatment, and can be part of a strategy to stop using nicotine right away or to reduce consumption with a view to quitting later. According to the opinion of the High Council of Public Health of 22 February 2016, ZYBAN and CHAMPIX can be prescribed as second-line medications for smoking cessation.

The electronic cigarette is not recommended to date as a smoking cessation aid, but can be a smoking cessation aid.

Hypnosis, cognitive and behavioral therapies, acupuncture are also used for withdrawal.

Auriculotherapy (ART) is based on the observation that treating specific points on the pinna improves some symptoms, relieves pain and anxiety. It is practiced in the context of Pain Assessment and Treatment Centers (PATC) where it is particularly effective on certain stubborn pains, in supportive care and in cancerology. It is also effective in general medicine where it provides an interesting non-drug therapeutic aid. It is also used in smoking cessation.

Auriculotherapy is taught in France within the framework of an inter-university diploma (Strasbourg- Paris XI). The doctors involved in this study have all been trained in this way and regularly use ART by integrating it into their practice within the Foch's PATC.

Cryo-auriculotherapy treatment (injection of nitrous oxide at -89°C) is a simple and powerful treatment since the effect of one session seems to last, depending on the indications, for about 1 to 4 weeks, thus reducing the number of sessions required.

We hypothesized that ART treatment by cryotherapy of specific points of the auricle could help smoking cessation.

This first proof-of-concept project, named StopAuric, is realized to validate our hypothesis on a population of motivated patients who will not use nicotine substitutes in order to measure the impact of cryo-ART alone.

It is a prospective, multicenter, controlled, single-blind, randomized study in 2 parallel groups.

Patients will be randomized into 2 groups :

* Experimental group "True Cryo-auriculotherapy": Patients will be treated with auriculotherapy with N2O (nitrogen) projection on specific smoking cessation points.
* "Sham" control group: the patients will be treated according to the same scheme as the experimental group with a technique without N2O (sham cryotherapy), but with the presence of the propellant gaz.

Responses to the Hospital Anxiety and Depression Scale (HADS), Patient Global Impression of Change questionnaire (PGIC) self-questionnaires, satisfaction VAS, possible weight gain, smoking consumption, and measurement of exhaled Carbon mOnoxide (CO) and urinary cotinine will be collected at one month.

Patients will be able to say whether or not they wish to continue the same treatment.

If this proof-of-concept study is positive regarding the interest of an ART session in smoking cessation, we planned to initiate a larger study (named Auriculo-TABAC) evaluating the value of a complete ART treatment program in smoking cessation.

This largest study will treat patients of the experimental arm with CryoAuriculotherapy over 3 sessions (D0, D30 and D60).

The expected effect of smoking cessation will be evaluated at 3 and 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Be of legal age
* Have an active smoking habit
* Wish to quit smoking and nicotine completely (VAS of motivation ≥ 7 on a scale of 0 to 10)
* Have signed a consent form;
* Be affiliated with a health insurance plan.

Exclusion Criteria:

* Contraindication to the use of auriculotherapy (lesion or infection of the auricle) by cryotherapy (skin healing disorder, risk of hypo or hyperpigmentation);
* Treatment with Varenicline (Champix®, etc...) or Bupropion hydrochloride (Zyban®, etc...) in progress; treatment with nicotine substitutes (patches, gum, nicotine e-cigarette)
* Treatment by auriculotherapy or acupuncture in this indication in the previous 12 months;
* Previous treatment with cryo-auriculotherapy;
* Having to start any new smoking cessation treatment that could interfere with the study: specific drug treatment (antidepressant, morphine, anticonvulsant) or complementary therapy (psychological or mind-body treatment);
* Difficulty complying with the treatment, questionnaire or study protocol;
* Being deprived of liberty or under guardianship.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2021-11-16 (Actual); Primary Completion 2023-10-23 (Actual); Study Completion 2023-10-23 (Actual)

PRIMARY OUTCOMES:
Confirmation that cryotherapy auriculotherapy is effective in the treatment of smoking cessation compared to a "sham" treatment (without N2O). | 1 month
  Percentage of patients who quit smoking at 1 month, judged on urine cotinine (value <50μg/l) between the 2 groups.

SECONDARY OUTCOMES:
Evaluation of the effect of auriculotherapy by cryotherapy on side effects of smoking cessation : stress | 1 Month
  Perceived Stress Scale will be used at the inclusion and at the one month follow-up visit to assess changes in the perceived stress by patient.
  The scale ranges from 0 to 10. 0 being the lowest stress level and 10 the highest.
Evaluation of the effect of auriculotherapy by cryotherapy on side effects of smoking cessation : anxiety and depression | 1 Month
  Hospital Anxiety and Depression questionnaire will be used at inclusion and at 1 month post-treatment.
  There are seven questions related to anxiety (total A) and seven others related to the depressive dimension (total D), allowing thus obtaining two scores (maximum score of each score = 21).
  Higher score indicates a certain symptomatology :
  7 or less: absence of symptoms 8 to 10: doubtful symptomatology 11 and more: certain symptomatology.
Evaluation of the effect of auriculotherapy by cryotherapy on side effects of smoking cessation : weight gain | 1 month
  Weight changes between the inclusion visit and the 1 month post-treatment visit will be assessed
Patient Global Impression of Change questionnaire (PGIC) used at the end of the follow-up. | 1 month
  This scale evaluates all aspects of patients' health and assesses if there has been an improvement or decline in clinical status with a seven-point single-item scale ranging from 'very much worse' to 'very much improved
Willingness of the patient to continue treatment | 1 month
  Patient will be asked at the end of the study if they want to pursue the treatment
Tolerance of cryotherapy auriculotherapy treatment. | 1 month
  The presence or absence of adverse events attributed to the treatment of auriculotherapy by the patient.

CONTACTS AND LOCATIONS:
Overall Officials: Mireille MICHEL-CHERQUI, MD, Principal Investigator — Hôpital Foch; Marc FISCHLER, MD PhD, Study Director — Hôpital Foch
Locations (3):
- France (3):
  - Espace Santé Simone Veil, Issy-les-Moulineaux, Hauts De Seine
  - Clinique de la Sauvegarde, Lyon, Rhône
  - Cabinet de l'Olivier, Montigny-le-Bretonneux, Yvelines

IPD SHARING:
Plan to Share IPD: No